CLINICAL TRIAL: NCT06612840
Title: An Open-label, Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics or Preliminary Efficacy and Antitumor Activity of GNC-077 Multi-specific Antibody Injection in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer and Other Solid Tumors
Brief Title: A Study of GNC-077 in Patients With Locally Advanced or Metastatic Non-small-cell Lung Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-077-101
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GNC-077 (Experimental): Participants receive GNC-077 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-077

INTERVENTIONS:
Drug: GNC-077 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter, dose-escalation and cohort expansion phase I clinical study to evaluate the safety, tolerability, pharmacokinetics characteristics or preliminary efficacy and antitumor activity in patients with Locally advanced or metastatic non-small cell lung cancer and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the informed consent form, voluntarily participate in and sign the informed consent form;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old (stage Ia); ≥18 years old (stage Ib);
4. Locally advanced or metastatic non-small cell lung cancer and other solid tumors;
5. Must have at least one measurable lesion that meets the RECIST v1.1 definition;
6. have archived primary or recurrent tumor tissue specimens that can be submitted for central review;
7. ECOG ≤1;
8. The expected survival time as judged by the investigators was ≥3 months;
9. Bone marrow function, renal function and liver function should meet the requirements;
10. Coagulation function: fibrinogen ≥1.5g/L; Activated partial thromboplastin time (APTT) ≤1.5×ULN; Prothrombin time (PT) ≤1.5×ULN;
11. Fertile female subjects or male subjects with fertile partners must use highly effective contraception from 7 days before the first dose until 12 weeks after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose;
12. Subjects were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
2. Patients with active infection requiring intravenous antibiotics who did not complete treatment within 1 week before enrollment;
3. Positive human immunodeficiency virus antibody, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
4. No reduction in toxicity from previous antineoplastic therapy to grade I as defined in CTCAE, version 5.0, or to the level specified in the inclusion criteria;
5. Patients at risk for active autoimmune disease or with a history of autoimmune disease may have central nervous system involvement;
6. Pulmonary disease defined as ≥ grade 3 according to NCI-CTCAE v5.0; A history of ILD requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis;
7. Patients with previous allogeneic hematopoietic stem cell transplantation or organ transplantation;
8. Had a history of severe cardiovascular and cerebrovascular diseases;
9. Patients had or had thrombotic events such as deep vein thrombosis, arterial thrombosis and pulmonary embolism within 6 months before screening;
10. Brain parenchymal metastases and/or meningeal metastases or spinal cord compression, excluding stable and asymptomatic brain parenchymal metastases;
11. Uncontrolled pleural effusion with clinical symptoms who were judged by the investigator to be ineligible for enrollment;
12. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
13. Who had participated in a clinical trial of an unmarketed drug within 4 weeks before the trial dose;
14. Had received a live vaccine within 4 weeks before the trial dose;
15. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ia: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-077 . The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-077.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-077.

SECONDARY OUTCOMES:
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of GNC-077 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of GNC-077 will be investigated.
AUC0-inf | Up to approximately 24 months
  AUC0-inf is defined as area under the concentration-time curve from 0 to inf.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of GNC-077 per unit of time will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of GNC-077 will be investigated.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-GNC-077 antibody (ADA) will be investigated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-077 to the first date of either disease progression or death, whichever occurs first.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PHD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China